CLINICAL TRIAL: NCT04603079
Title: A Randomized Control Trial to Change Nurse Leadership in Maintaining Minimum Service Delivery Standards for Hospital Infection Control in the Era of COVID-19
Brief Title: Nurse Leadership for Hospital Infection Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Forman Christian College, Pakistan (Other)
Collaborators: King Edward Medical University (Other)
Responsible Party: Principal Investigator, Sara Rizvi Jafree, Assistant Professor, Department of Sociology, Forman Christian College, Pakistan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NurseLeadership
Record Dates: First submitted 2020-10-19; First posted 2020-10-26 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Nurse's Role; Infection
Keywords: Randomized Control Trial; Nurse leadership; Hospital Infection Control; COVID-19
MeSH Terms: conditions — Infections; COVID-19 | interventions — Methods

STUDY DESIGN:
Intervention Model Description: A total of 200 nurses will be sampled. A 100 nurses each will be randomly assigned to the control and experiment group each.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Currently practicing nurses who will receive intervention (Experimental): An intervention for COVID-19 preventive protocols will be delivered to the nurses in the experiment group.
  Interventions: Behavioral: Intervention for COVID-19 preventive protocols
- Currently practicing nurses who will not receive intervention (No Intervention): No intervention for COVID-19 preventive protocols will be delivered to the nurses in the control group.

INTERVENTIONS:
Behavioral: Intervention for COVID-19 preventive protocols — The intervention will comprise (A) digital communication of written material and (B) monthly online training and discussion through skype and zoom, to allow for physical demonstrations, Q&A and sharing of challenges. The five specific areas covered in the intervention for COVID-19 preventive protocols will include: (1) PPE fitting, (2) PPE removal, (3) hand hygiene, (4) cleaning, disinfection and sterilization, and (5) nurse uniform sterilization.
  Arms: Currently practicing nurses who will receive intervention

SUMMARY:
The aim is to deliver an intervention to promote nurse leadership and decision-making in the hospital setting, by providing them with training for maintaining minimum service delivery standards for hospital infection control with respect to COVID-19; but also other infectious disease burden management.

DETAILED DESCRIPTION:
Nurses are frontline practitioners in the fight against COVID-19. Empowering nurses through training for infection prevention for COVID-19 is an essential step to facilitate nurse leadership and safety in the hospital. There is immense reliance on nurses with regard to patient safety, yet very little effort is made to invest in interventions for their leadership roles in developing countries, including Pakistan. In this study the aim is to deliver an intervention for COVID-19 preventive protocols to nurses and assess the impact of the intervention through a pre and post-test survey. A total of 200 nurses will be sampled. A 100 nurses each will be part of the control and experiment group each.

The data will be analyzed using SPSS. Pre and post test results will be presented using descriptive data and bivariate regression will be used to present higher odds of confidence in preventive and awareness literacy for COVID-19 in nurses after intervention delivery. Through this research the aim is to improve nurse leadership in maintaining minimum service delivery standards for hospital infection control with respect to COVID-19; but also other infectious disease burden management.

ELIGIBILITY:
Inclusion Criteria:

* The selection criteria will be all currently working staff nurses.

Exclusion Criteria:

* Student nurses or nurses not part of clinical rounds.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 344 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Core competencies in nurses for infection control and prevention (Min and Sil 2014) | 3 months
  It will consist of 44 questions for core competencies of infection control and prevention, including 10 constructs of: (1) Identification of infectious disease processes, (2) Surveillance and epidemiologic investigations, (3) Preventing/controlling the transmission of infectious agents, (4) Employee/occupational health, (5) Management and communication planning, (6) Quality/performance improvement and patient safety, and (7) Education and research education, (8) Confidence with training and awareness for identification and implementation for COVID-19 prevention and control strategies, (9) confidence in training and awareness, and (10) satisfaction with workplace support. It is a five-point Likert-type scale (strongly agree - agree - neutral - disagree - strongly disagree). The highest value of the scale is 6 and the lowest value is 1; with 6 points showing strong agreement with the item statement (E.g. Q1. Can you differentiate between other infections and COVID-19).

CONTACTS AND LOCATIONS:
Locations (1):
- Online sampling of nurses from public and private hospitals (confidential data), Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
All SPSS data files will be made publicly available. No names of participants will be shared, only participant codes.
Supporting Information: Study Protocol, SAP, ICF